CLINICAL TRIAL: NCT06827496
Title: Initial Oral Antibiotics for Bone and Joint Infections in Children: A Prospective Nationwide Real-world Effectiveness Study in Denmark
Brief Title: Initial Oral Antibiotics for Bone and Joint Infections in Children
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Innovation Fund Denmark (Individual)
Responsible Party: Principal Investigator, Ulrikka Nygaard, Ass Professor, Consultant, PhD, MD, MPhil, Rigshospitalet, Denmark
Other Study IDs: P-2029-29; 0176-00020B (Other Grant/Funding Number: Innovation Fund Denmark)
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Osteomyelitis Acute; Septic Arthritis; Bone Infection; Joint Infection; Bone and Joint Infection
Keywords: Bone and joint infections; Children; Oral antibiotics; Osteomyelitis
MeSH Terms: conditions — Arthritis, Infectious; Osteomyelitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Plasma and serum samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children and adolescents with bone and joint infections treated with initial oral antibiotics: Patients with uncomplicated bone and joint infections treated with initial oral antibiotics.
  According to Danish Nationwide Guidelines (initiated in 2024), initial oral antibiotics are recommended to patients with no risk factors for complicated disease. Risk factors include for complicated disease include:
  1. Severe illness or sepsis
  2. Rapid symptom progression
  3. Pronounced symptoms, including severe pain
  4. Pronounced soft tissue involvement
  5. Foreign material or post-surgical infection
  6. Infection with a resistent or rare pathogen, e.g., Salmonella or MRSA
  7. Severe comorbidity, including immunodeficiency
  Patients who have received intravenous antibiotic therapy for less than 24 h before oral antibiotics will be included
  Interventions: Drug: Oral antibiotic treatment

INTERVENTIONS:
Drug: Oral antibiotic treatment — Initial antibiotics:
  Below 5 years: High-dose amoxicillin-clavulanate (8:1 ratio; 100/12.5 mg/kg/day in 3 doses) until clinical improvement and decrease in CRP, followed by dose reduction (4:1 ratio) to 50/12.5 mg/kg/day in 3 doses).
  5 years and above: High-dose anti-staphylococcal penicillin (200 mg/kg/day in 4 doses) until clinical improvement and decrease in CRP, with dose reduction (100 mg/kg/day in 4 doses) after clinical improvement
  Treatment duration of follow-up therapy (after initial high-dose antibiotics): One week for uncomplicated joint infections, three weeks for bone infections, and four weeks for spondylodiscitis

SUMMARY:
Initial oral antibiotic treatment for children and adolescents with uncomplicated bone and joint infections (BJI) has been found non-inferior to initial IV antibiotics in one randomized controlled trial (RCT). The real-world effectiveness of initial oral antibiotics for children and adolescents with BJI is unclear.

This nationwide, prospective, multicenter, real-world cohort study aims to compare the effectiveness and safety of initial oral antibiotic treatment for children and adolescents with uncomplicated BJI in a real-world setting with those who received initial oral antibiotics in our RCT.

DETAILED DESCRIPTION:
Background:

Initial oral antibiotic treatment for children and adolescents with uncomplicated BJI has been found non-inferior to initial IV antibiotics in one randomized controlled trial (RCT) from Denmark. The real-world effectiveness of initial oral antibiotics for children and adolescents with BJI is unclear. In Denmark, initial oral antibiotics were allowed in nationwide guidelines for children and adolescents aged 3 months to 17 years with uncomplicated BJI from 2024.

Aim:

We aim to compare the effectiveness and safety of initial oral antibiotics for children and adolescents with uncomplicated BJI in a real-world setting with those who received initial oral antibiotics in our RCT.

Study design:

Nationwide, prospective, multicenter, real-world cohort study.

Patients:

100 children and adolescents aged 3 months to 17 years with uncomplicated BJI treated with initial oral antibiotics at one of the 18 Pediatric Departments in Denmark from 2024 to 2026. Uncomplicated BJI is defined by the absence of impaired general condition or signs of sepsis, rapidly progressing or severe symptoms, pronounced soft tissue involvement, prosthetic material, resistant pathogens, and severe comorbidities. Patients who have received intravenous antibiotic therapy for less than 24 h before oral antibiotics will be included.

Control patients are 98 patients who received initial oral antibiotics for uncomplicated BJI as part of a Danish RCT conducted between 2020 and 2023.

Methods:

All children and adolescents treated for BJI will be prospectively enrolled. Designated co-investigators in the 18 Danish pediatric departments will ensure prospective, national inclusion. Follow-up assessments will be conducted after three, six, 12 month. The three-month follow-up will include a clinical examination to ensure full recovery. The six and 12-month follow-up will be conducted via a structured telephone interview and/or a clinical evaluation.

All study data will be securely collected and managed in an online database.

Outcomes:

The primary outcome is sequelae after 6 months, defined as any atypical mobility or function of the affected bone or joint.

Secondary outcomes are suspicion of treatment failure within 28 days, full recovery after initiation of treatment, recurrent infection within 6 months, and sequelae after 12 months and 5 years.

Safety outcomes are surgical intervention and severe complications during antibiotic treatment.

We will calculate the risk difference sequelae between the real-world and RCT cohorts using exact unconditional two-sided 95% confidence interval.

ELIGIBILITY:
Children and adolescents aged 3 months to 17 years with uncomplicated bone and joint infections treated with initial oral antibiotics.

According to Danish Nationwide Guidelines (initiated in 2024), initial oral antibiotics are recommended to patients with no risk factors for complicated disease. Risk factors include for complicated disease include:

1. Severe illness or sepsis
2. Rapid symptom progression
3. Pronounced symptoms, including severe pain
4. Pronounced soft tissue involvement
5. Foreign material or post-surgical infection
6. Infection with a resistent or rare pathogen, e.g., Salmonella or MRSA
7. Severe comorbidity, including immunodeficiency

Patients who have received intravenous antibiotic therapy for less than 24 h before oral antibiotics will be included

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 3 months to 17 years with uncomplicated bone and joint infections treated with initial oral antibioticsbetween 15th of November 2024 and 15th of November 2026
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Clinical sequelae at 6 months | 6 months after end of treatment [4-9 months]
  Clinical sequelae is defined as any abnormal mobility or function of the affected bone or joint.
  Clinical sequelae will be evaluated through a structured medical telephone interview at 6 months with a parent or a guardian (or the patient, if adolescent, along with the parent). If the medical interview raises any concerns about abnormal mobility or function of the affected bone or joint, or if the patient is scheduled for a clinical consultation, clinical sequelae will be evaluated by a clinical examination performed by a pediatrician or an orthopedic surgeon.

SECONDARY OUTCOMES:
Suspicion of treatment failure within 28 days | 28 days after initiation of treatment
  Change of antibiotic therapy due to suspicion of treatment treatment failure or slow recovery, such as persistent fever for more than 3 days, iincrease in C-reactive protein after 4 days, or absence of clinical improvement within 5 days of treatment initiation.
Full recovery after initiation of treatment | Within 3 months after initiation of treatment (0-4 months)
  Full recovery is defined as absence of clinical features of the affected bone or joint. Assessment made by a pediatrician or orthopedic surgeon.
Recurrent infection within 6 months | 6 months after the end of treatment
  Recurrence of symptoms and signs requiring readministration of antibiotics after initial recovery and cessation of antibiotic treatment.
Clinical sequelae at 12 months | 12 months after the end of treatment [9-16 months]
  Clinical sequelae is defined as any abnormal mobility or function of the affected bone or joint.
  Clinical sequelae will be evaluated through a structured medical telephone interview at 12 months with a parent or a guardian (or the patient, if adolescent, along with the parent). If the medical interview raises any concerns about abnormal mobility or function of the affected bone or joint, or if the patient is scheduled for a clinical consultation, clinical sequelae will be evaluated by a clinical examination performed by a pediatrician or an orthopedic surgeon.
Sequelae at 5 years | 5 years after the end of treatment [4-6 years]
  Sequelae is defined as any abnormal mobility or function of the affected bone or joint.
  The child is deemed to have no long-term clinical sequelae if there are no hospital contacts for atypical mobility or function of the affected bone or joint and if he/she is still registered as residing in Denmark (defined as 'lost to follow-up' if no longer residing in Denmark)

OTHER OUTCOMES:
Safety outcome 1: Surgical intervention | 28 days after initiation of treatment
  Surgical intervention during antibiotic treatment excluding diagnostic interventions, such as diagnostic bone biopsy or diagnostic joint aspiration with or without lavage.
Safety outcome 2: Severe complications during antibiotic treatment | 28 days after initiation of treatment
  Severe complications during antibiotic treatment, e.g. need for intensive care, septic shock, organ failure, pyomyositis, endocarditis, deep venous thrombosis.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrikka Nygaard, Ass Professor, PhD, MD, MPhil, Study Chair — Copenhagen University Hospital, Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen Ø, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bybeck Nielsen A, Borch L, Damkjaer M, Glenthoj JP, Hartling U, Hoffmann TU, Holm M, Helleskov Rasmussen A, Schmidt LS, Schmiegelow K, Stensballe LG, Nygaard U; Local Investigators. Oral-only antibiotics for bone and joint infections in children: study protocol for a nationwide randomised open-label non-inferiority trial. BMJ Open. 2023 Jun 1;13(6):e072622. doi: 10.1136/bmjopen-2023-072622. PMID 37263683